CLINICAL TRIAL: NCT00390624
Title: Prevention Of Nephrotoxicity Following Allogeneic Bone Marrow Transplantation Using Urodilatin (Ularitide,Atrial Natriuretic Peptide) and Mannitol.
Brief Title: Prevention Of Nephrotoxicity Following Bone Marrow Transplantation Using Urodilatin and Mannitol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rocky Mountain Cancer Centers (Other)
Collaborators: University of Colorado, Denver (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RMBMT-123
Record Dates: First submitted 2006-10-19; First posted 2006-10-20 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-05

CONDITIONS: Renal Dysfunction; Acute Renal Failure; Mortality
Keywords: Urodilatin; Mannitol; Acute Kidney Failure
MeSH Terms: conditions — Renal Insufficiency; Acute Kidney Injury | interventions — Ularitide; Atrial Natriuretic Factor; Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: URODILATIN (ULARITIDE, ATRIAL NATRIURETIC PEPTIDE)
Drug: MANNITOL

SUMMARY:
The purpose of the study is to combine Urodilatin (ANP analogue), which will increase glomerular filtration rate (GFR), and mannitol, which will increase the rate of urinary flow and solute excretion. We intend to treat twenty consecutive allogeneic bone marrow transplant patients in a phase II study comparing results with historical controls.

We hypothesize that the incidence of renal dysfunction, ARF and thus mortality in allogeneic bone marrow transplantation can be significantly reduced by the use of protective agents Urodilatin and mannitol. We feel that this combination is best administered prior to and during the first two weeks of treatment when patients encounter immunosuppressive agents and the onset of early transplantation complications.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Presence of malignancy or hematological disease whose treatment will be allogeneic stem cell transplant and high-dose conditioning therapy.
* Adequate baseline evaluation: adequate renal function (creatinine clearance > 60 ml/min); Adequate hepatic function (SGOT, SGPT, bilirubin and alkaline phosphatase < 1.5 times normal); adequate cardiac function (MUGA showing a left ventricular ejection at rest > 45%); adequate pulmonary function (DCLO > 60%).

Exclusion Criteria:

* Known hypersensitivity to ANP or mannitol
* Congestive heart failure
* Previous bone marrow transplant
* BP less than 90 mm systolic or less than 60 mm Hg diastolic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2003-07; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Renal function will be assessed for first 30 days after transplantation for the primary endpoint.
The primary endpoints will be a comparison of the grades of renal dysfunction, incidence of ARF requiring dialysis, and overall survival

SECONDARY OUTCOMES:
Patient will be followed at 3 month intervals for the first year and then yearly for life.

CONTACTS AND LOCATIONS:
Overall Officials: Chirag R Parikh, MD, PhD, Principal Investigator — Yale School of Medicine (Nephrology)
Locations (1):
- Rocky Mountain Cancer Centers 1800 Williams Street, Suite 200, Denver, Colorado, United States

REFERENCES:
- [Background] Zager RA, O'Quigley J, Zager BK, Alpers CE, Shulman HM, Gamelin LM, Stewart P, Thomas ED. Acute renal failure following bone marrow transplantation: a retrospective study of 272 patients. Am J Kidney Dis. 1989 Mar;13(3):210-6. doi: 10.1016/s0272-6386(89)80054-x. PMID 2645771
- [Background] Gruss E, Bernis C, Tomas JF, Garcia-Canton C, Figuera A, Motellon JL, Paraiso V, Traver JA, Fernandez-Ranada JM. Acute renal failure in patients following bone marrow transplantation: prevalence, risk factors and outcome. Am J Nephrol. 1995;15(6):473-9. doi: 10.1159/000168889. PMID 8546168
- [Background] Letourneau I, Dorval M, Belanger R, Legare M, Fortier L, Leblanc M. Acute renal failure in bone marrow transplant patients admitted to the intensive care unit. Nephron. 2002 Apr;90(4):408-12. doi: 10.1159/000054728. PMID 11961399
- [Background] Merouani A, Shpall EJ, Jones RB, Archer PG, Schrier RW. Renal function in high dose chemotherapy and autologous hematopoietic cell support treatment for breast cancer. Kidney Int. 1996 Sep;50(3):1026-31. doi: 10.1038/ki.1996.405. PMID 8872980
- [Background] Parikh CR, McSweeney PA, Korular D, Ecder T, Merouani A, Taylor J, Slat-Vasquez V, Shpall EJ, Jones RB, Bearman SI, Schrier RW. Renal dysfunction in allogeneic hematopoietic cell transplantation. Kidney Int. 2002 Aug;62(2):566-73. doi: 10.1046/j.1523-1755.2002.00455.x. PMID 12110019